CLINICAL TRIAL: NCT04957745
Title: Monocular Visual Confusion for Field Expansion
Brief Title: Understanding Visual Confusion Using Stereoscopic Displays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Jaehyun Jung, Assistant Professor, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021P001757; R01EY031777 (NIH)
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Diplopia; Binocular Vision Suppression; Binocular; Fusion, With Defective Stereopsis; Monocular Diplopia
Keywords: Visual confusion; Rivalry; Head mounted display; Stereoscopic displays; Binocular vision
MeSH Terms: conditions — Diplopia

STUDY DESIGN:
Intervention Model Description: All participants in the group will see all three interventions (peripheral targets in three visual confusion conditions) in a randomized order. In this study design, each participant will serve as their own control, and the order of the interventions will be randomized to account for potential carryover or ordering effects. There will be no comparison or control group. The outcome will be compared through a within-subject analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual confusion (Experimental): Participants viewed peripheral targets in three different visual confusion conditions (three interventions): binocular visual confusion (unilateral opaque target), unilateral monocular visual confusion (unilateral see-through target), and bilateral monocular visual confusion (bilateral see-through target). Each intervention was presented twice in a randomized order, resulting in a total of six trials. During each trial, a peripheral target was presented in front of a forward-moving background for one minute. Participants were instructed to hold down the controller button while the target was visible and release it when a third or more of the target disappeared. After each trial, participants could take a brief break before the next trial in a different visual confusion condition was presented in a randomized order.
  Interventions: Behavioral: Binocular visual confusion (unilateral opaque); Behavioral: Unilateral monocular visual confusion (unilateral see-through); Behavioral: Bilateral monocular visual confusion (bilateral see-through)

INTERVENTIONS:
Behavioral: Binocular visual confusion (unilateral opaque) — The peripheral target was a horizontally drifting grating measuring 10° by 10°, with a spatial frequency of 1 cycle per degree and a temporal frequency of 3 Hz, and located at 10° above the fixation.
  For the binocular visual confusion condition, the non-transparent (opaque) peripheral target will be displayed on only one eye (unilateral opaque display).
Behavioral: Unilateral monocular visual confusion (unilateral see-through) — The peripheral target was a horizontally drifting grating measuring 10° by 10°, with a spatial frequency of 1 cycle per degree and a temporal frequency of 3 Hz, and located at 10° above the fixation.
  For the unilateral monocular visual confusion condition, the half-transparent peripheral target will be displayed on only one eye (unilateral see-through display).
Behavioral: Bilateral monocular visual confusion (bilateral see-through) — The peripheral target was a horizontally drifting grating measuring 10° by 10°, with a spatial frequency of 1 cycle per degree and a temporal frequency of 3 Hz, and located at 10° above the fixation.
  For bilateral monocular visual confusion condition, the half-transparent peripheral target will be displayed on both eyes (bilateral see-through display).

SUMMARY:
In this research study we want to test how people understand a visual scene when the same image is presented to both the eyes, but portions of these images are altered in terms of contrast, depth or in some cases motion.

ELIGIBILITY:
Inclusion Criteria:

* Better than 20/40 visual acuity in the worse eye
* No restrictions of the peripheral visual field: (at least 60 degrees vertically and 40 degrees horizontally)
* At least 14 years of age (no upper age limit)
* Able to give voluntary, informed consent
* Able to understand English
* Binocular vision parameters within normal limits (Stereopsis ≤ 100 arc sec on any stereo test)

Exclusion criteria:

* Patients with any physical or mental disabilities, including cognitive dysfunction, balance problems, or other deficits that could impair their ability to respond to the stimuli presented in this study will be excluded
* Being unable to complete sessions lasting 2-3 hours

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JaeHyun Jung, Principal Investigator — Schepens Eye Research Institute
Locations (1):
- Schepens Eye Research Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 participants were recruited and screened for eligibility and all of them met the inclusion criteria.
Pre-assignment Details: 13 participants were recruited and screened for eligibility and all of them met the inclusion criteria.
Period: Overall Study
Arm/Group | Visual Confusion
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Visual Confusion: The study participants will respond to various visual confusion stimuli presented on a stereoscopic display designed to simulate binocular/monocular visual confusions
  Visual confusion: We will show peripheral target images on a background motion in a stereoscopic display. For the binocular visual confusion condition, the target peripheral image will be displayed on only one eye. For unilateral and bilateral monocular visual confusion conditions, the half-transparent peripheral image will be displayed on only one eye and both eyes, respectively.
Arm/Group | Visual Confusion
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.46 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-hispanic | 5
  Asian/Non-hispanic | 8
Region of Enrollment [Number; unit: participants]
  United States | 13
Visual acuity [Mean (Standard Deviation); unit: Snellen fraction (20/X)] — The visual acuity test is used to determine the smallest letters that a participant can read on a standardized chart (Snellen chart) held 20 feet away. A Snellen fraction of 20/20 indicates normal vision, where the smallest line of letters on the chart can be read from 20 feet away. For example, 20/40 (worse than normal) vision can see a letter clearly at 20 feet that normal vision could see clearly at 40 feet, while 20/10 (better than normal) vision can see a letter clearly at 20 feet that normal vision could see clearly at 10 feet. We measured visual acuity with both eyes open.
  Snellen fraction (20/X) | 19.38 (4.21)
Stereo-acuity [Mean (Standard Deviation); unit: arcseconds] — Stereo acuity refers to the smallest detectable depth difference that can be perceived through binocular vision. It is measured in terms of the angular difference in arcseconds, with smaller values indicating better acuity. The random dot stereogram is commonly used to measure stereoacuity within the range of 20 to 400 arcseconds. In this test, participants are asked to identify which of three circles appears to float forward or seems "different" from the others. If the participant's stereoacuity is better than the target value, they will be able to discern the differences.
  arcseconds | 27.7 (9.28)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Total Viewing Time That Peripheral Target is Perceived
Description: (Total time the peripheral target in the visual confusion condition was visible) / (total viewing time (=1 min))
Time Frame: Approximately 1-2 sessions to finish total 6 trials, up to 2 hours for each session, any time within the 4month study period
Population: Each subject observed two trials in each visual confusion condition. There were three visual confusion conditions, so each subject participated in 6 trials. Since 13 subjects participated, the total number of trials analyzed was 78 trials (6 * 13). For each visual confusion condition, 26 trials were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Units Other Than Participants: Trials
Groups:
- Visual Confusion: Participants viewed peripheral targets in three different visual confusion conditions (three interventions) - Binocular visual confusion (unilateral opaque target), Unilateral monocular visual confusion (unilateral see-through target), and Bilateral monocular visual confusion (bilateral see-through target) - twice in a randomized order, resulting in a total of six trials.
  During each trial, the peripheral target in a different visual confusion in front of a forward-moving background was presented to the participant for 1 minute. Participants were instructed to hold down the controller button while the target was visible and release it when a third or more of the target disappeared.
  After each trial, participants could take a brief break (e.g., blinking eye) before the next trial in a different visual confusion condition was presented in a randomized order.
Arm/Group | Visual Confusion
Number analyzed (Participants) | 13
Number analyzed (Trials) | 78
Percentage of Time
  Binocular visual confusion (unilateral opaque target) | 73.56 (17)
  Unilateral monocular visual confusion (unilateral see-through target) | 59.64 (25.42)
  Bilateral monocular visual confusion (bilateral see-through target) | 87.81 (13.85)
Statistical Analysis 1: Comparison: Visual Confusion; Effect of visual confusion conditions (binocular, unilateral monocular, and bilateral monocular visual confusions) on "Percentage of Total Viewing Time Peripheral Target is Perceived" is analyzed by repeated measure (within-subject) ANOVA. The test was performed with a significance level of 0.05; Test type: Other; p < 0.01, ANOVA — Null hypothesis is that there is no difference in "Percentage of Total Viewing Time that Peripheral Target is Perceived" across visual confusion conditions

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 months, for all three interventions
Description: All participants who saw at least one intervention (peripheral target in any visual confusion condition) were asked to report when they experienced any potential other adverse events (i.e., dizziness, motion sickness, and nausea), but there were no reported other adverse events.
Arm/Group | Visual Confusion
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT04957745/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT04957745/ICF_001.pdf